CLINICAL TRIAL: NCT07025213
Title: Metabolic Effect of a Physical Activity and Dietary Intervention, and Its Association With Musculoskeletal Changes, in Endometrial Cancer Patients Eligible for Staging Surgery, Compared to Patients Not Receiving the Physical Activity Intervention. A Pilot Study.
Brief Title: Metabolic Effect of Exercise and Diet in Endometrial Cancer Patients Eligible for Staging Surgery.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cancerología (Other Government)
Responsible Party: Principal Investigator, Lucely Cetina Pérez, Dr., National Institute of Cancerología
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: (024/046/ICI)(CEI/041/24)
Record Dates: First submitted 2025-05-22; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Endometrial Cancer
Keywords: excercise; muscle mass and strength; Metabolism changes; inflammation biomarkers; quality of life; surgical complication
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Diet; Exercise

STUDY DESIGN:
Intervention Model Description: Open-label, two-arm pilot study in adult women diagnosed with endometrial cancer and candidates for staging surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet. (Active Comparator): This group will only receive recommendations to follow an anti-inflammatory diet.
  Interventions: Other: Diet.
- Diet and exercise. (Experimental): The intervention group will receive both dietary and exercise interventions.
  Interventions: Other: Diet and exercise.

INTERVENTIONS:
Other: Diet and exercise. — The intervention group will receive recommendations to follow an anti-inflammatory diet. In addition, they will be instructed to increase their level of physical activity and will be asked to attend the institute to carry out a supervised exercise routine.
  Arms: Diet and exercise.
Other: Diet. — The comparison group will be instructed to follow the anti-inflammatory diet intervention only.
  Arms: Diet.

SUMMARY:
Background:

Endometrial cancer is one of the diseases linked to obesity in women. In Mexico, about 7.6 women out of every 100,000 are diagnosed with this type of cancer, and nearly three-quarters of these women have obesity. Many women with endometrial cancer also have a condition called sarcopenic obesity, where muscle loss happens but might not be easy to identify. Researchers believe that certain molecules in the blood could help identify the health of muscles. Exercise helps muscles stay strong and healthy by affecting these molecules. For women with cancer, staying active can help maintain muscle mass, which is important for better recovery and health outcomes. This project focuses on an exercise program for women with locally advanced endometrial cancer who will be treated surgically at the National Cancer Institute of Mexico (INCan).

What We Think Will Happen:

Women with endometrial cancer who participate in a program combining physical activity and healthy eating will gain more muscle strength and function compared to those who don't exercise. We expect these changes to be connected to healthier levels of certain molecules in the blood, showing less muscle breakdown and less inflammation. We also believe these women will have better control of blood sugar and fats.

Our Main Goal:

To find out how physical activity and diet affect muscle health and metabolism in women with endometrial cancer, and to compare these changes to women who don't participate in the exercise program.

How We Will Do It:

We will measure molecules related to muscle health in the blood. We will also assess muscle size, strength, and how well the muscles work. Then, we will look for connections between these muscle changes and the blood molecules. We want to see if improvements in muscle are linked to better recovery from surgery and better health outcomes. If so, these blood molecules might help doctors monitor muscle health. We hope that the exercise program will help women recover better and improve their quality of life.

How We Will Analyze the Data:

We will describe the data we collect and compare the group that exercises to the group that doesn't. We will use statistics to see if the differences are meaningful. We will also analyze the relationship between muscle health and blood markers. Advanced methods will help us identify which molecules and measurements best explain the changes seen. The results will be carefully reviewed using specialized software.

What We Hope to Find:

We aim to show that blood tests can help identify muscle health and how it improves with exercise. This could lead to earlier detection of muscle loss and better management through exercise programs. Ultimately, this work hopes to improve the health and well-being of women facing endometrial cancer.

DETAILED DESCRIPTION:
What is Endometrial Cancer (EC)?

* EC is a cancer that starts in the lining of the uterus.
* The number of cases worldwide, including Mexico, has been rising steadily over the past decades.
* Most cases are found early (stage I), and there are two main types:

Type I (most common): linked to hormones like estrogen, usually has a better outlook.

-Type II: less common and not related to estrogen.

What Increases the Risk of EC?

* Being overweight or obese is a major risk factor because fat tissue produces estrogen, which can fuel the cancer.
* Other risks include diabetes, high blood pressure, and lack of physical activity.
* Obesity causes chronic inflammation in the body, creating an environment that supports cancer growth.
* What is Sarcopenia and Sarcopenic Obesity?
* Sarcopenia means losing muscle strength and mass, often due to aging or diseases like cancer.
* Sarcopenic obesity is when someone has both excess fat and low muscle, which is linked to worse health outcomes in cancer patients.
* In EC patients, sarcopenia and obesity together can make treatment harder and lower survival rates.

How Does Obesity Affect EC Treatment?

* Obesity increases surgical risks and can limit treatment options.
* Patients with good muscle mass before surgery tend to recover better and live longer.
* Comorbidities (like diabetes or heart disease) common in obesity can complicate cancer treatment.
* Role of Physical Activity
* Exercise is very beneficial for people with EC, obesity, and sarcopenia.
* Aerobic (cardio) exercise helps reduce fat, especially around organs.
* Resistance (strength) training helps build muscle mass and improve strength.
* Exercise can reduce inflammation, improve metabolism, and enhance quality of life.
* For cancer patients, staying active helps manage side effects, improve treatment tolerance, and reduce fatigue.

Importance of Diet

* A healthy diet rich in fruits, vegetables, whole grains, healthy fats, and protein supports weight management and muscle health.
* Avoid diets high in sugar, unhealthy fats, and processed foods, which contribute to obesity and inflammation.
* Nutritional support should start at diagnosis to improve treatment outcomes and overall health.

What Patients and Families Should Know

* Maintaining a healthy weight and staying physically active can reduce the risk of EC and improve outcomes if diagnosed.
* Muscle strength and nutrition are very important during cancer treatment.
* Work with healthcare providers to develop a plan that includes diet, physical activity, and medical treatment tailored to individual needs.
* Early detection and timely treatment improve prognosis.

What Healthcare Providers Should Know

* Screen for obesity, diabetes, hypertension, and sarcopenia in patients with or at risk for EC.
* Counsel patients on the benefits of physical activity and healthy eating.
* Consider multidisciplinary care involving nutritionists, physical therapists, and oncologists.
* Monitor muscle mass and function as part of cancer care to improve surgical and treatment outcomes.
* Tailor treatment plans considering the patient's physical condition and comorbidities.

General Objective:

To evaluate the metabolic effect of a physical activity and dietary intervention in patients with endometrial cancer who are candidates for staging surgery, and its association with musculoskeletal changes, in comparison with a control group of patients who do not receive the physical activity intervention.

Hypothesis Patients with endometrial cancer who engage in physical activity and follow a dietary intervention will show an increase in skeletal muscle mass, strength, and function compared to women who do not engage in physical activity. This change will be associated with a serum amino acid profile, an increase in molecules related to anabolism, a decrease in those related to catabolism, and changes in the cytokine profile indicating a trend toward reduced inflammation. Additionally, women who undergo the physical activity intervention will show improvements in glucose and lipid metabolism compared to those who do not engage in physical activity.

ELIGIBILITY:
Inclusion Criteria:

1. -Ability to understand the nature of the study and provide written informed consent.
2. -Women aged over 18 and under 65 years.
3. -Availability to attend exercise sessions.
4. -Willingness and ability to comply with scheduled visits, the proposed nutritional algorithm, treatment plan, and laboratory tests.
5. -Histologically confirmed diagnosis of endometrioid-type endometrial cancer by biopsy.
6. -Normal electrocardiogram (ECG) result.
7. -No prior oncological treatment.
8. -Body mass index (BMI) greater than 20 kg/m².
9. -Availability of a computed tomography (CT) scan.
10. -Candidates for staging surgery.

Exclusion Criteria:

1. -Patients with advanced clinical stage or stage IVB disease (according to FIGO 2018 criteria).
2. -Patients with a prior or concurrent malignancy, except non-melanoma skin cancer.
3. -Patients with uncontrolled systemic arterial hypertension.
4. -Patients with renal dysfunction (eGFR ≤ 60 mL/min/1.73 m²).
5. -Patients with uncontrolled psychiatric disorders, including claustrophobia.
6. -Patients with concurrent infections.
7. -Patients with autoimmune disease.
8. -Patients with neuromuscular disease.
9. -Contraindications to physical exercise.
10. -Vulnerable situations (e.g., homelessness preventing adherence to diet, or incarceration).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in serum tyrosine concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum histidine concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum lysine concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum phenylalanine concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum glutamic acid concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum methionine concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum aspartic acid concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum proline concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum serine concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum threonine concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum isoleucine concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum valine concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum leucine concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum glycine concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum cystine concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum alanine concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum IL-6 concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum IL-10 concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum TGF-betha concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum TNF-alpha concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum creatine kinase concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum irisin concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum decorin concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in serum musclin concentration after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks
Changes in total blood cholesterol after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks.
Changes in blood LDL cholesterol after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks.
Changes in blood HDL cholesterol after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks.
Changes in blood triglycerides after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks.
Changes in blood glucose after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks.
Changes in insulin after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks.
Changes in glycosylated hemoglobin after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks.
Changes in muscle mass after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks.
Changes in hand strength after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks.
Changes in physical function after the physical activity plus diet intervention, compared to patients receiving diet only. | From enrollment to the end of treatment at 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Denisse Castro Eguiluz, PhD, Principal Investigator — Ministry of Science, Humanities and Technology (SECIHTI)-National Cancer Institute.
Locations (1):
- Instituto Nacional de Cancerología, México, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No